CLINICAL TRIAL: NCT04370535
Title: Evaluation of PMA-Zeolite-Clinoptilolite Effects on the Dysbiosis and Inflammation in Patients With Uncontrolled Crohn Disease
Brief Title: PMA-Zeolite-Clinoptilolite Effects in Crohn Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ciim Plus, d.o.o. (Industry)
Collaborators: University of Rijeka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: crohn-disease ver. 1.3_17
Record Dates: First submitted 2018-05-04; First posted 2020-05-01 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: The pilot-study is a randomized, placebo-controlled and double blinded study. The 4 subject-groups are consisting of group A and B with healthy subjects (A and B are divided into a placebo-group and into a PMA-zeolite- group) and group C and D which are subjects suffering from CD (C and D are divided into a placebo-group and into a PMA-zeolite- group). No washout phase is planned, but if food-supplements are taken this will be protocolled. The diagnostics will be performed through the defined parameters at defined time-points.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group + cellulose (Group A) (Placebo Comparator): healthy subjects (control group) receive placebo (cellulose) as powder
  Interventions: Device: cellulose
- Control group + PMA-zeolite(Group B) (Active Comparator): healthy subjects (control group) receive PMA-zeolite as powder
  Interventions: Device: PMA-zeolite
- UCD-group + Cellulose (Group C) (Placebo Comparator): subjects with uncontrolled Crohn disease (UCD group) receive placebo (cellulose) as powder
  Interventions: Device: cellulose
- UCD-group + PMA-zeolite (Group D) (Active Comparator): subjects with uncontrolled Crohn disease receive PMA-zeolite as powder
  Interventions: Device: PMA-zeolite

INTERVENTIONS:
Device: cellulose — The subjects of group A and group C receive boxes containing placebo for supplementation for a total of 12 weeks.
  Arms: Control group + cellulose (Group A); UCD-group + Cellulose (Group C)
Device: PMA-zeolite — The subjects of group B and group D receive boxes containing PMA-zeolite for supplementation for a total of 12 weeks.
  Arms: Control group + PMA-zeolite(Group B); UCD-group + PMA-zeolite (Group D)

SUMMARY:
This pilot study aims to evaluate the safety and efficacy of PMA-zeolite when used in patients with uncontrolled CD (Crohn´s disease). The effect of the PMA-zeolite will be compared between a control-group (healthy volunteers) receiving either PMA-zeolite or placebo and the test-group (suffering from uncontrolled CD) and receiving either PMA-zeolite or placebo. In addition, this pilot-study should furthermore provide indications for the effect-size in order to estimate an effect for an eventual further human trial.

DETAILED DESCRIPTION:
Background of the study Crohn´s disease (CD) is a chronic progressive destructive disease. Approximately one-fifth of adult and paediatric patients already have evidence of a structuring or penetrating intestinal complications at diagnosis. Despite decades of research, the aetiology of CD remains unknown. Disease treatments include a variety of approaches like dietary changes and immunosuppressive anti-TNFa antibodies as well as ancillary antibiotic therapy. Another interesting and promising approach in this context might be the supplementation of the certified medical device PMA-(Panaceo micro activation)-zeolite (a specific natural zeolite-clinoptilolite) due to its properties documented through many studies. In particular, the promising clinical results from a randomized controlled trial (RCT) with PMA-zeolite need to be highlighted. The strengthening/ supporting of the intestinal wall integrity in healthy subjects suffering from intestinal problems was measured in this RCT and is claimed as intended main action of the PMA-zeolite. Based on these results the application of PMA-zeolite is an interesting and promising approach in patients with uncontrolled CD.

Hypothesis In the present trial, it is being tested if supplementing PMA-zeolite can lead to an improvement of the defined markers and parameters (reduction of local and systemic inflammation, changes of the microbiota in the gut, positive detoxifying effect and general improvement of quality of life) in patients with uncontrolled CD compared to a healthy test-group.

Aims This pilot study aims to evaluate the safety and efficacy of PMA-zeolite when used in patients with uncontrolled CD. The effect of the PMA-zeolite will be compared between a control-group (healthy volunteers) receiving either PMA-zeolite or placebo and the test-group (suffering from uncontrolled CD) and receiving either PMA-zeolite or placebo. In addition, this pilot-study should furthermore provide indications for the effect-size in order to estimate an effect for an eventual further human trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (at least 18 years old) for first two groups (A,B), homogenous starting group in age (30-60Y) and sex (m/f )

  o The health-status will be confirmed through anamnesis.
* Groups C and D will include patients with confirmed Crohn's disease that are treated with standard therapy and despite of treatment do not achieve the appropriate disease remission. Patients with the intermediate type of disease will be also included in groups C and D.

  * Diagnosis has to be confirmed with a biopsy of the intestine and histological exam.
  * Degree of disease will be assessed by Harvey-Bradshaw Index (HBI). For evaluation of quality BDQ questionnaire will be used. For the assessment of disease activity ordinary laboratory measurements will be performed (CBC, basic biochemical parameters, CRP), and calprotectin from chairs. Colonoscopy must be done in the last six months prior to inclusion of patients in the research protocol. Gastrointestinal system degree of impairment will not have influence on inclusion criteria and patients with histological intermediate type of disease will be included as well.
* Signed informed consent as per usual recommendations in vigour in the Republic of Slovenia.

Exclusion Criteria:

* Signs of acute bacterial infection (fever >38°C, nausea, vomiting).
* Other chronic disease (cancer, renal disease, neuro-degenerative, metabolic disorders, diabetic).
* Pregnancy or breastfeeding
* Food supplements** **NOTE: Food supplements: if taken regularly this should be continued also during the study and documented - otherwise a wash - out - phase would be necessary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Zonulin concentration in stool (ng/ml) | 0(baseline) and after 12 weeks
  As the intestinal wall permeability is linked to several conditions, such as the Crohn Disease it is hypothesized that a change of Zonulin (biomarker for permeability of intestinal wall) is detectable with/without supplementation of the study-substance.
  Measurement: stool stool sample (by ELISA kit) Standard Value for Zonulin: < 55 ng/ml .

SECONDARY OUTCOMES:
Bacterial diversity in the marbus crohn patients | 0(baseline) and after 12 weeks
  bactieria of assessment: Lactobacillus, Escherichia, bifidobacteria
  Measurement: stool sample (16S RNA sequencing on stool sampling)

OTHER OUTCOMES:
Changes of blood parameters | 0(baseline) and after 12 weeks
  Blood samples for measurement of definied parameters:
  * Ni: 0,6-3,8 µg/L
  * Al: < 7,0 µg/L
  * Na: 3100,0 - 3350,0 mg/L
  * K: 140,0 - 200,0 mg/L
  * Mg: 17,0-23,0 mg/L
  * Ca: 89,0-101,0 mg/L
  * Se: 70,0-150,0 µg/L
  * Zn: 660,0-1100,0 µg/L
  * Cu: 750,0-1450,0 µg/L
  * Fe: M: 550,0-1600,0 µg/L
  * F: 400,0-1550,0 µg/L DAO (Standard Value > 10 U/ml ), ammonia - µmol/l,histamine (ng/ml), Measurement of sedimentation, blood count, electrolytes, urea, liver-parameters, creatinine and other
Rate of Safety and tolerability | 0(baseline) and after 12 weeks
  Rate of tolerability and safety levels of minerals and metals

CONTACTS AND LOCATIONS:
Overall Officials: Krešimir Pavelić, PhD, M.D., Principal Investigator — Juraj Dobrila University of Pula
Locations (3):
- Slovenia (3):
  - University Clinical Centre Ljubljana, Ljubljana
  - Medical Thermal Centre Fontana, Maribor
  - Slovenj Gradec General Hospital, Slovenj Gradec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraljevic Pavelic S, Saftic Martinovic L, Simovic Medica J, Zuvic M, Perdija Z, Krpan D, Eisenwagen S, Orct T, Pavelic K. Clinical Evaluation of a Defined Zeolite-Clinoptilolite Supplementation Effect on the Selected Blood Parameters of Patients. Front Med (Lausanne). 2022 May 27;9:851782. doi: 10.3389/fmed.2022.851782. eCollection 2022. PMID 35712111